CLINICAL TRIAL: NCT00253708
Title: Body-Based Complementary Therapies for Patients With Cancer
Brief Title: Massage Therapy in Treating the Symptoms of Patients With Locally Advanced or Metastatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Russell Phillips, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2003P000299; CDR0000445117 (Registry Identifier: PDQ (Physician Data Query)); R21CA098487 (NIH)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2017-08-07 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-06

CONDITIONS: Cancer
Keywords: depression; nausea and vomiting; pain; psychosocial effects of cancer and its treatment; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; extensive stage small cell lung cancer; stage III gastric cancer; stage III esophageal cancer; localized unresectable adult primary liver cancer; stage III colon cancer; stage IV renal cell cancer; stage IV bladder cancer; stage IV prostate cancer; stage IV breast cancer; stage IV ovarian epithelial cancer; advanced adult primary liver cancer; stage IV melanoma; stage IV ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; recurrent small cell lung cancer; recurrent adult primary liver cancer; recurrent colon cancer; recurrent esophageal cancer; recurrent gastric cancer; recurrent non-small cell lung cancer; recurrent bladder cancer; recurrent breast cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent prostate cancer; recurrent renal cell cancer; recurrent melanoma
MeSH Terms: conditions — Neoplasms; Depression; Nausea; Vomiting; Pain; Carcinoma, Non-Small-Cell Lung; Stomach Neoplasms; Esophageal Neoplasms; Colonic Neoplasms; Carcinoma, Renal Cell; Urinary Bladder Neoplasms; Prostatic Neoplasms; Breast Neoplasms; Carcinoma, Ovarian Epithelial; Melanoma; Small Cell Lung Carcinoma; Carcinoma, Hepatocellular | interventions — Massage; Analgesia; Psychiatric Rehabilitation

STUDY DESIGN:
Intervention Model Description: The study was designed to assess the feasibility and effectiveness of massage for patients with cancer-related pain
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- massage (Experimental): Patients received 3 massage therapy visits from massage therapists in initial week with a duration of 15-45 minutes.NOTE: Intervention 'management of therapy complications' has not been included in any Arm/Group Descriptions.
  Patients were intended to receive pain therapy, psychosocial assessment and care, and quality-of-life assessment
  Interventions: Procedure: management of therapy complications; Procedure: massage therapy; Procedure: pain therapy; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment
- no-touch control (Active Comparator): Patients received 3 no-touch therapy visits from massage therapists who provided no-touch without healing intention.Patients were intended to receive pain therapy, psychosocial assessment and care, and quality-of-life assessment
  Interventions: Procedure: management of therapy complications; Procedure: massage therapy; Procedure: pain therapy; Procedure: psychosocial assessment and care; Procedure: quality-of-life assessment
- Usual care (No Intervention): Patients did not receive visits from massage therapists. Patients were intended to receive pain therapy, psychosocial assessment and care, and quality-of-life assessment

INTERVENTIONS:
Procedure: management of therapy complications
  Arms: massage; no-touch control
Procedure: massage therapy
  Arms: massage; no-touch control
Procedure: pain therapy
  Arms: massage; no-touch control
Procedure: psychosocial assessment and care
  Arms: massage; no-touch control
Procedure: quality-of-life assessment
  Arms: massage; no-touch control

SUMMARY:
RATIONALE: Massage therapy may help relieve symptoms associated with cancer. It is not yet known which type of massage therapy is more effective in treating the symptoms of patients with cancer.

PURPOSE: This randomized clinical trial is studying different types of massage therapy to compare how well they work in treating the symptoms of patients with locally advanced or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the safety and tolerated dose (i.e., duration, techniques, and degree of pressure) of professional massage therapy vs professional simple presence (no touch) massage therapy vs usual care followed by caregiver massage therapy vs usual care in patients with locally advanced or metastatic cancer.
* Correlate these therapies with pain, anxiety, depression, nausea, and shortness of breath in these patients.
* Correlate these therapies with patient quality of life and caregiver anxiety and depression.
* Determine the feasibility of teaching family caregivers how to provide massage therapy and the subsequent use of massage by the caregivers.
* Determine the effects of caregiver massage therapy on patients and caregivers.
* Determine the feasibility and acceptability among patients and massage therapists of a simple presence (no touch) massage therapy control group.

OUTLINE: This is a randomized, controlled, pilot study. Patients are randomized to 1 of 3 treatment arms.

* Arm I (professional massage therapy): Hospitalized patients are offered massage therapy by a licensed massage therapist for 15-45 minutes once daily for the duration of their hospital stay. Outpatient oncology clinic patients are offered home-based massage therapy by a licensed massage therapist for 15-45 minutes once daily for 3 days.
* Arm II (usual care): Patients receive usual care for symptom management.
* Arm III (professional simple presence [no touch] massage therapy): Hospitalized patients are offered simple presence (no touch) massage therapy comprising a room visit by a licensed massage therapist who places his/her hands 12 inches over the patient without direct touch for 15-45 minutes. Treatment is offered once daily for the duration of the hospital stay. Outpatient oncology clinic patients are offered home-based simple presence (no touch) massage therapy by a licensed massage therapist for 15-45 minutes once daily for 3 days.

All patients are then randomized (a second time) to 1 of 2 treatment arms.

* Arm I (caregiver massage therapy): Previously hospitalized patients are offered home-based caregiver massage therapy for 1 month. Outpatient oncology clinic patients are offered home-based caregiver massage therapy for 3 weeks.
* Arm II (usual care): Patients receive usual care for symptom management. Hospitalized patients complete a questionnaire addressing symptoms, quality of life, satisfaction with symptom control, and time spent up or out of bed once daily on days 1-5, every 3 days while in the hospital, and then at 1 week, 2 weeks, and 1 month after discharge from the hospital. Outpatient oncology clinic patients complete a similar telephone questionnaire at baseline, 1 week, and then at 1 month.

PROJECTED ACCRUAL: Approximately 100 patients will be accrued for this study.

ELIGIBILITY:
Inclusion criteria:

* Solid cancer with evidence of metastases
* Receiving treatment at Beth Israel Deaconess Medical Center (BIDMC)
* Must reside ≤ 25 miles from BIDMC

Exclusion criteria:

* Patient to sick to be interviewed
* Absence of severe symptoms
* Participating in another trial
* Language barrier
* MD does not provide permission
* Expired prior to consent process

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2004-12-01 (Actual); Primary Completion 2013-01-01 (Actual); Study Completion 2013-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell S. Phillips, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toth M, Marcantonio ER, Davis RB, Walton T, Kahn JR, Phillips RS. Massage therapy for patients with metastatic cancer: a pilot randomized controlled trial. J Altern Complement Med. 2013 Jul;19(7):650-6. doi: 10.1089/acm.2012.0466. Epub 2013 Jan 31. PMID 23368724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Using oncology clinic electronic database, eligible patients were selected based on their clinical diagnosis (solid cancer with evidence of metastases) and whether they lived within 25 miles of the hospital. Patients were told that the authors were conducting a study of nonpharmacologic treatments intended to improve symptom management.
Groups:
- Touch Intervention (Massage Therapy): Patients received three visits by the professional massage therapists over the first week after the enrollment. Massage treatments were scheduled based on patient preferences, and the duration was between 15 and 45 minutes; both the duration and the amount of pressure was modified depending on patient comfort. A limited scope of practice was provided to the massage therapists that specified the allowed and disallowed massage modalities and techniques. Allowed techniques were both Swedish and non-Swedish massage including gliding/effleurage, gentle kneading/petrissage, compression, gentle stretching, rocking, light myofascial release, active and/or passive range of motion, warm or cool applications, and use of acupressure points as well as craniosacral holds thought to have calming and centering effects. No forms of friction, deep-tissue massage, or bodywork forms that required movement by the patients were allowed.
- No Touch Intervention (Control): The authors wanted to separate out the effect of interacting with a massage therapist from massage itself, so the therapists performed no-touch control interventions, which had no healing intention. Although most of the therapists had experience with energy healing, the therapists were trained to avoid ''healing intention'' in the no-touch group by using distraction if necessary, created by counting backwards. For the no-touch control intervention, therapists were instructed to be with the patients between 15 and 45 minutes, depending on the patient's tolerance, and to hold their hands about 12 inches over the patient's body. In the usual-care control group, patients completed the same questionnaires but did not receive any visits from the massage therapists.
- Usual Care (Control): Patients did not receive visits from massage therapists. Patients were intended to receive pain therapy, psychosocial assessment and care, and quality-of-life assessment
Period: Overall Study
Arm/Group | Touch Intervention (Massage Therapy) | No Touch Intervention (Control) | Usual Care (Control)
Started | 20 | 10 | 9
Completed | 20 | 10 | 8
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Massage: Patients received 3 massage therapy visits from massage therapists in initial week with a duration of 15-45 minutes.NOTE: Intervention 'management of therapy complications' has not been included in any Arm/Group Descriptions.
  Patients were intended to receive pain therapy, psychosocial assessment and care, and quality-of-life assessment
  management of therapy complications
  massage therapy
  pain therapy
  psychosocial assessment and care
  quality-of-life assessment
- No-touch Control: Patients received 3 no-touch therapy visits from massage therapists who provided no-touch without healing intention.Patients were intended to receive pain therapy, psychosocial assessment and care, and quality-of-life assessment
  management of therapy complications
  massage therapy
  pain therapy
  psychosocial assessment and care
  quality-of-life assessment
- Total: Total of all reporting groups
Arm/Group | Massage | No-touch Control | Usual Care | Total
Number analyzed (Participants) | 20 | 10 | 9 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (12) | 54.9 (10) | 55.6 (9) | 55.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 6 | 32
  Male | 3 | 1 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 0 | 1
  White | 19 | 9 | 8 | 36
Marital status: Married, Other [Count of Participants; unit: Participants]
  Married | 13 | 6 | 8 | 27
  Other | 7 | 4 | 1 | 12
Living alone [Count of Participants; unit: Participants] | 3 | 2 | 0 | 5
Not admitted to hospital in the last 12 months [Count of Participants; unit: Participants] | 8 | 6 | 4 | 18
Education: College grad or more [Count of Participants; unit: Participants] | 10 | 6 | 5 | 21
Employment: full-time or part-time [Count of Participants; unit: Participants] | 5 | 5 | 4 | 14
Household income: Not available/refused/don't know, <$50,000, >$50,000 [Count of Participants; unit: Participants]
  Not available/refused/Don't know | 3 | 3 | 1 | 7
  <$50,000 | 4 | 2 | 1 | 7
  >$50,000 | 13 | 5 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: 0=no pain to 10=most severe pain
Time Frame: From baseline to 1 week and from baseline to one month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | 0 [-2 to 1] | 0 [-1 to 2] | 0 [-3 to 2]
  1 month | 0 [-1 to 0] | 0 [-1.5 to 0] | -2 [-2 to -1]

2. Primary Outcome: Anxiety
Description: 0=no anxiety to 10=most severe anxiety
Time Frame: From baseline to 1 week and from baseline to 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | 0 [-3 to 0] | 0 [-3 to 0] | 0 [-2 to 0]
  1 month | 0 [-2 to 0] | 0 [-1.5 to 1] | 0 [-3 to 0]

3. Primary Outcome: Alertness
Description: 0=not at all alert to 10=most alert
Time Frame: From baseline to 1 week and from baseline to 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | 0 [0 to 0] | 0 [-0.5 to 0] | 1 [0 to 2]
  1 month | 0 [-1 to 0] | 0 [-1.5 to 0] | 0 [0 to 1]

4. Secondary Outcome: Quality of Life: Physical Well-being
Description: Physical well-being over past 2 days (0= physically terrible to 10= physically well)
Time Frame: From baseline to 1 week and from baseline to 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | 1 [0 to 2] | -0.5 [-2 to 0.5] | 0 [-2 to 0]
  1 month | 0 [-1 to 1] | 0 [-3.5 to 0] | 0 [0 to 0]

5. Secondary Outcome: Quality of Life: Psychological Well-being
Description: Psychological well-being over past 2 days (depressed, nervous/worried, sad, terrified of future) (0= always/extremely to 10= never/not at all; in other words: 0=negative/worst to 10= positive/best)
Time Frame: From baseline to 1 week and from baseline to 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | 1.125 [0 to 2] | 0.25 [-0.5 to 2] | 0 [0 to 0.75]
  1 month | -0.125 [-0.5 to 0.5] | 0.25 [-1.25 to 1.5] | 0.75 [0 to 1.5]

6. Secondary Outcome: Quality of Life: McGill Total
Description: Quality of Life (McGill Total); Mean of five sub-measures (but not overall) (0 = negative to 10 = positive)
Time Frame: From baseline to 1 week and from baseline to 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | 0.45 [0 to 1.23] | 0 [-0.66 to 0.28] | 0 [-0.57 to 0]
  1 month | 0 [-0.42 to 0.3] | -0.18 [-1.29 to 0.13] | 0 [0 to 0.58]

7. Secondary Outcome: Sleep
Description: Sleep (Richards-Campbell) 0 = best sleep to 50 = worst sleep
Time Frame: From baseline to 1 week and from baseline to 1 month
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Massage | No-touch Control | Usual Care
Number analyzed (Participants) | 20 | 10 | 9
units on a scale
  1 week | -3.5 [-9 to 0] | 0 [-7 to 9] | -0.5 [-4 to 1]
  1 month | -4 [-12 to 0] | 0 [-12 to 10] | 0 [-15 to 12]

ADVERSE EVENTS:
Time Frame: From baseline to 1 month
Description: There were no study-related adverse events.
Arm/Group | Massage | No-touch Control | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10 | 1/9
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/20 | 0/10 | 0/9

LIMITATIONS AND CAVEATS:
Small sample size limited statistical power. Pre-post intervention data collection was not blinded. Patient bias in massage group. Heterogeneity in type and stage of cancer may have resulted in variation of the effects of the interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes